CLINICAL TRIAL: NCT05548738
Title: The Efficacy of Ultrasound and Fluoroscopy Guided Caudal Epidural Prolotherapy Versus Steroids for Chronic Pain Management in Failed Back Surgery Syndrome
Brief Title: Caudal Epidural Prolotherapy Versus Steroids in Failed Back Surgery Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Ahmed Shehab, MD, Lecturer in Anaesthesia and Surgical ICU department, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0201626
Record Dates: First submitted 2022-09-14; First posted 2022-09-21 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Chronic Pain Syndrome
Keywords: caudal epidural; prolotherapy; steroids; failed back surgery
MeSH Terms: interventions — Steroids; Prolotherapy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor) double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Steroid group (Group S) (Active Comparator): This group will receive ultrasound and fluoroscopy-guided caudal epidural steroid injection
  Interventions: Drug: medthylprednisolone
- Prolotherapy group (Group P) (Experimental): This group will receive ultrasound and fluoroscopy-guided caudal epidural prolotherapy injection
  Interventions: Drug: prolotherapy

INTERVENTIONS:
Drug: medthylprednisolone — a type of steroids injected in epidural space
  Other Names: steroids
  Arms: Steroid group (Group S)
Drug: prolotherapy — a type of hypertonic glucose
  Other Names: dextrose 10%
  Arms: Prolotherapy group (Group P)

SUMMARY:
This study will be held on patients with failed back surgery syndrome, the investigators are comparing prolotherapy and steroids injections in caudal epidural space to relieve the pain

DETAILED DESCRIPTION:
This study is a prospective double blinded randomized controlled study. It will be held on patients with failed back surgery syndrome aged between 20 and 70 years old, one group will receive ultrasound and fluoroscopy-guided injection of prolotherapy in caudal epidural space while the other group will receive ultrasound and fluoroscopy-guided injection of steroids in the caudal epidural space 40 patients will be included in each group

ELIGIBILITY:
Inclusion Criteria:

1. patients diagnosed with failed back surgery syndrome, having chronic pain for more than 3 months by a detailed assessment including medical history and examination
2. patients having positive radiological (MRI) findings of spinal nerve roots being irritated or compressed after having surgery for one of many conditions including: lumbar disc herniation, spinal canal stenosis, osteophytes, spodylolithesis or foramen stenosis
3. patients whom another surgery is not indicated

Exclusion Criteria:

1. patient refusal
2. pregnancy
3. systemic infection or infection at the site of injection
4. patients on anticoagulation
5. immunocompromised patients as uncontrolled diabetes, osteoporosis as a contraindication for steroid injection
6. patients with renal impairment or on dialysis
7. acute disc prolapse as it requires immediate surgery
8. opioid use
9. concurrent significant depressive illness, inflammatory of joint disease.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Assessing in both groups the Visual analogue scale from 0-10 where 0 indicates no pain and 10 indicates maximum pain | 2 weeks
  A decrease in VAS score after 2 weeks by 50 percent or more from pre-injection level is considered successful

SECONDARY OUTCOMES:
the level reached by the injectate | at time of injection
  by using fluoroscopy guidance
assessing the patient satisfaction by a the short assessment of patient satisfaction score (SAPS) from 0 to 28 where 0 is so dissatisfied and 28 means very satisfied | 6 months
  assess the satisfaction of the patients
further change in visual analogue scale | 2 weeks till 6 months
  in the next follow up periods
recording the number of patients who encountered any complications and treating them accordingly | 6 months
  such as pain, allergy, swelling at the site of injection, nerve injury, elevated blood sugar level, nausea and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed S shehab, Principal Investigator — Alexandria University
Locations (1):
- Ahmed S. Shehab, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
there is a plan to make individual participant data (IPD) collected in this study, including data dictionaries, available to other researchers
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After study ends upon request
Access Criteria: Accessible through the web site

REFERENCES:
- [Result] Maniquis-Smigel L, Reeves KD, Rosen HJ, Lyftogt J, Graham-Coleman C, Cheng AL, Rabago D. Analgesic Effect and Potential Cumulative Benefit from Caudal Epidural D5W in Consecutive Participants with Chronic Low-Back and Buttock/Leg Pain. J Altern Complement Med. 2018 Dec;24(12):1189-1196. doi: 10.1089/acm.2018.0085. Epub 2018 Jun 8. PMID 29883193